CLINICAL TRIAL: NCT04849390
Title: A Randomized, Placebo-controlled, Double-blind Trial Evaluating the Efficacy, Tolerability and Safety of ESO-101 in Adult Patients With Active Eosinophilic Esophagitis
Brief Title: A Study to Investigate the Efficacy and Tolerability of ESO-101 in Patients With Eosinophilic Esophagitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EsoCap AG (Industry)
Collaborators: FGK Clinical Research GmbH (Industry); FGK Representative Service B.V. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACESO; 2020-000082-16 (EudraCT Number)
Record Dates: First submitted 2021-04-02; First posted 2021-04-19 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The placebo will be identical to the test product in terms of appearance, constitution of inactive ingredients, packaging, labeling and administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESO-101 (Experimental): Oral use of 1 hard gelatin capsule (800 μg)
  Interventions: Drug: ESO-101
- Placebo (Placebo Comparator): Oral use of 1 hard gelatin capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ESO-101 — Daily administration in the evening at bedtime for 28 days
  Other Names: Mometasone furoate (800 μg)
  Arms: ESO-101
Drug: Placebo — Daily administration in the evening at bedtime for 28 days
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled, double-blind trial to evaluate the efficacy, tolerability, and safety of ESO-101 in adult patients with active eosinophilic esophagitis (EoE). Patients will be screened at 2 visits (Visit 1 and Visit 2) during which their eligibility will be assessed based on endoscopy-independent criteria (Visit 1) and based on the histologic assessment of esophageal biopsy samples taken during the screening endoscopy (Visit 2). Eligible patients will be randomized 2:1 to once-daily treatment with ESO-101 or placebo and treated for 28 days starting on Day 0. Further clinic visits will be performed at Day 14 (Visit 4) and Day 28 (Visit 5, end of treatment) to assess the efficacy, tolerability, and safety. In addition, a safety follow-up call will be scheduled 2 weeks after the end of treatment (Day 42, Visit 6).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18-70 years;
2. Confirmed clinicopathological diagnosis of EoE (eosinophilic esophagitis);
3. Active and symptomatic EoE, defined as:

   1. peak eosinophil count ≥15 eosinophils/high-powered field (hpf) at 2 levels of the esophagus at the screening endoscopy (Visit 2) as measured in a total of 6 hpfs derived from 6 biopsies, 2 each from the proximal, mid, and distal segment of the esophagus;
   2. either a dysphagia or odynophagia severity sore of ≥4 on a 11-point numeric rating scale for ≥1 day during the 7 days before Screening (Visit 1);
4. Written informed consent;
5. Willingness and ability to comply with the protocol for the duration of the trial;
6. Negative pregnancy test at Screening (Visit 1) and Day 0 (Visit 3) in women of childbearing potential (i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy);
7. Women of childbearing potential must be willing to use (for a least 3 monthly cycles before the screening endoscopy [Visit 2] and until 4 weeks after the last intake of IMP) a highly effective method of contraception or birth control (failure rate less than 1% per year when used consistently and correctly). Reliable methods for this trial are:

   1. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal);
   2. progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable);
   3. intrauterine device or intrauterine hormone-releasing system;
   4. bilateral tubal occlusion;
   5. a vasectomized sexual partner;
   6. sexual abstinence (only accepted as true abstinence when this is in line with the preferred and usual lifestyle of the patient; periodic abstinence [e.g. calendar, ovulation, symptothermal, post-ovulation methods, and withdrawal] is not an acceptable method of contraception).

Exclusion Criteria:

1. Women who are pregnant, lactating, possibly pregnant or planning a pregnancy during the trial period;
2. Current or past (within the last 3 months) alcohol or drug abuse;
3. Initiation of a diet-modifying food restriction within 4 weeks before the screening endoscopy (Visit 2) until EOT (end of treatment);
4. Use of systemic corticosteroids or biologic immunomodulators within 3 months before the screening endoscopy (Visit 2) until the EOT;
5. History of non-response to treatment of EoE with topical corticosteroid drugs (defined as no improvement of clinical symptoms of EoE after a minimum of 4 weeks corticosteroid therapy used at appropriate doses according to the investigator's judgment) or requirement of cessation of corticosteroid therapy for EoE treatment due to oral candidiasis or systemic corticosteroid side effects;
6. Use of corticosteroids for treatment of EoE within 4 weeks before the screening endoscopy (Visit 2) until the EOT;
7. Use of inhalable (pulmonary or nasal) corticosteroids within 4 weeks before the screening endoscopy (Visit 2) until the EOT;
8. Asthma requiring corticosteroid therapy in the seasonal allergy period according to the investigator's judgment based on anamnesis until the EOT;
9. Change in proton pump inhibitor (PPI) dosing regimen within 4 weeks before the screening endoscopy (Visit 2) until the EOT;
10. Use of systemic leukotriene receptor antagonists, immunosuppressant therapy, or chronic oral or systemic anticoagulants (such as coumarin derivates, novel oral and subcutaneous anticoagulants) within 2 weeks before Screening (Visit 1) until the EOT;
11. Unable to swallow a test tablet of about the size of the IMP capsule used in the trial;
12. History of diabetes mellitus;
13. Other severe comorbid condition, concurrent medication, or other issue that renders the patient unsuitable to participate in the trial in the judgment of the investigator, including but not limited to: comorbid condition with an estimated life expectancy of ≤12 months, dialysis, severe pulmonary (requiring home oxygen, uncontrolled chronic obstructive pulmonary disease Gold III/IV) or cardiovascular conditions (heart failure New York Heart Association III and IV, uncontrolled hypertension systolic blood pressure by repeated measurement >180mmHg);
14. History of cancer (except non-melanoma skin cancer, or carcinoma in situ of cervix) or treatment with anticancer therapy (chemotherapy, immunotherapy, radiotherapy, hormone therapy for cancer treatment, targeted therapy or gene therapy) within 12 months before Screening (Visit 1) until the EOT;
15. Known intolerability or hypersensitivity to mometasone furoate or any of the IMP excipients (e.g. bovine gelatin, polyvinyl alcohol, polyvinyl acetate, glycerol, sorbitol);
16. Systemic autoimmune disorders or any condition requiring immunosuppression (e.g. methotrexate, cyclosporine, interferon alpha, tumor necrosis factor alpha inhibitors, antibodies to immunoglobulin E) within 3 months before Screening (Visit 1);
17. Mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the trial or presence of any condition that impacts compliance with the trial procedures;
18. Use of any investigational or non-registered product (medicinal product or medical device) within 4 weeks before the screening endoscopy (Visit 2) until the EOT;
19. Employee at the trial center, spouse, partner or child of investigators or sub-investigators or employee of the sponsor.
20. History of or active eosinophilic gastroenteritis and colitis, inflammatory bowel disease, celiac disease, oral or esophageal mucosal infection of any kind, and esophageal varices;
21. Gastroesophageal reflux disease with Los Angeles Grade B or higher, or erosive esophagitis Grade 2 or above;
22. Presence of Barrett's esophagus with a maximum length of ≥3 cm with intestinal metaplasia or dysplasia, peptic stricture, achalasia, significant hiatal hernia >3 cm, esophageal scleroderma, or diagnosis of Lichen planus;
23. Emergency endoscopy for bolus impaction within 2 weeks before Screening (Visit 1);
24. Any mouth or dental condition that prevents normal eating;
25. History of (dilation within the previous 8 weeks) or current severe endoscopic structural abnormality in esophagus (e.g. high-grade stenosis where an 8-10 mm endoscope cannot pass without dilatation at the screening endoscopy [Visit 2]);
26. Diagnosed liver cirrhosis or portal hypertension;
27. History of upper gastrointestinal bleeding within 8 weeks before Screening (Visit 1);
28. Known allergy to β-lactoglobulin (cow milk protein).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2023-10-09 (Actual)

PRIMARY OUTCOMES:
Absolute change in peak eosinophil count from Baseline to end of treatment | From Baseline (Visit 2) to end of treatment (Visit 5 = 4-7 weeks after Visit 2)
  The processing and analysis of biopsy samples taken at Visit 2 and end of treatment (Visit 5) will be performed blinded at a central laboratory according to a laboratory manual. At both visits, 6 biopsy samples will be taken, 2 each from the proximal, mid, and distal segment of the esophagus. Histology results of the biopsies at Visit 2 will be considered baseline values. For the peak number of eosinophils, hematoxylin and eosin stained esophageal biopsy specimen will be assessed and the high-powered fields with the highest density of eosinophils will be counted.

SECONDARY OUTCOMES:
Proportion of patients with histological remission, defined as the reduction of peak eosinophil count in all esophageal samples to <15 eosinophils/hpf at end of treatment, overall and determined differentially in each of the 3 esophageal segments | From Baseline (Visit 2) to end of treatment (Visit 5 = 4-7 weeks after Visit 2)
  Biopsy samples will be taken at Visit 2 and end of treatment (Visit 5). At both visits, 6 biopsy samples will be taken, 2 each from the proximal, mid, and distal segment of the esophagus. Histology results of the biopsies at Visit 2 will be considered baseline values. For the peak number of eosinophils, hematoxylin and eosin stained esophageal biopsy specimen will be assessed and the high-powered fields (hpfs) with the highest density of eosinophils will be counted.
Proportion of patients with a peak eosinophil count in all esophageal samples of <6 eosinophils/hpf at end of treatment, overall and determined differentially in each of the 3 esophageal segments | End of treatment (Visit 5 = day 28)
  Biopsy samples will be taken at Visit 2 and end of treatment (Visit 5). At both visits, 6 biopsy samples will be taken, 2 each from the proximal, mid, and distal segment of the esophagus. Histology results of the biopsies at Visit 2 will be considered baseline values. For the peak number of eosinophils, hematoxylin and eosin stained esophageal biopsy specimen will be assessed and the high-powered fields (hpfs) with the highest density of eosinophils will be counted.
Proportion of patients with an improvement in the dysphagia severity score from Baseline to end of treatment | From Baseline (Visit 3) to end of treatment (Visit 5 = 28 days after Visit 3)
  Patients will rate the dysphagia severity score daily on a 11-point NRS (numeric rating scale): 0 = 'no symptoms' to 10 = 'worst possible symptoms'. At Visit 3 (Day 0) and Visit 5 (end of treatment), the worst severity scores out of the 7 days preceding the respective visit will be used for the assessment. The score assessed at Visit 3 (Day 0) at the center before IMP intake will serve as baseline score. Patients will additionally assess the severity score of the actual day in the patient diary daily after IMP intake starting on Day 0.
Absolute change in mean eosinophil count from Baseline to end of treatment | From Baseline (Visit 2) to end of treatment (Visit 5 = 4-7 weeks after Visit 2)
  The processing and analysis of biopsy samples taken at Visit 2 and end of treatment (Visit 5) will be performed blinded at a central laboratory according to a laboratory manual. At both visits, 6 biopsy samples will be taken, 2 each from the proximal, mid, and distal segment of the esophagus. Histology results of the biopsies at Visit 2 will be considered baseline values. For the peak number of eosinophils, hematoxylin and eosin stained esophageal biopsy specimen will be assessed and the high-powered fields with the highest density of eosinophils will be counted.
Relative change in mean eosinophil count from Baseline to end of treatment | From Baseline (Visit 2) to end of treatment (Visit 5 = 4-7 weeks after Visit 2)
  The processing and analysis of biopsy samples taken at Visit 2 and end of treatment (Visit 5) will be performed blinded at a central laboratory according to a laboratory manual. At both visits, 6 biopsy samples will be taken, 2 each from the proximal, mid, and distal segment of the esophagus. Histology results of the biopsies at Visit 2 will be considered baseline values. For the peak number of eosinophils, hematoxylin and eosin stained esophageal biopsy specimen will be assessed and the high-powered fields with the highest density of eosinophils will be counted.
Proportion of patients with a relative reduction in peak eosinophil count of ≥30 percent from Baseline to end of treatment | From Baseline (Visit 2) to end of treatment (Visit 5 = 4-7 weeks after Visit 2)
  The processing and analysis of biopsy samples taken at Visit 2 and end of treatment (Visit 5) will be performed blinded at a central laboratory according to a laboratory manual. At both visits, 6 biopsy samples will be taken, 2 each from the proximal, mid, and distal segment of the esophagus. Histology results of the biopsies at Visit 2 will be considered baseline values. For the peak number of eosinophils, hematoxylin and eosin stained esophageal biopsy specimen will be assessed and the high-powered fields with the highest density of eosinophils will be counted.
Proportion of patients with a relative reduction in peak eosinophil count of ≥50 percent from Baseline to end of treatment | From Baseline (Visit 2) to end of treatment (Visit 5 = 4-7 weeks after Visit 2)
  The processing and analysis of biopsy samples taken at Visit 2 and end of treatment (Visit 5) will be performed blinded at a central laboratory according to a laboratory manual. At both visits, 6 biopsy samples will be taken, 2 each from the proximal, mid, and distal segment of the esophagus. Histology results of the biopsies at Visit 2 will be considered baseline values. For the peak number of eosinophils, hematoxylin and eosin stained esophageal biopsy specimen will be assessed and the high-powered fields with the highest density of eosinophils will be counted.
Proportion of patients with a relative reduction in peak eosinophil count of ≥75 percent from Baseline to end of treatment | From Baseline (Visit 2) to end of treatment (Visit 5 = 4-7 weeks after Visit 2)
  The processing and analysis of biopsy samples taken at Visit 2 and end of treatment (Visit 5) will be performed blinded at a central laboratory according to a laboratory manual. At both visits, 6 biopsy samples will be taken, 2 each from the proximal, mid, and distal segment of the esophagus. Histology results of the biopsies at Visit 2 will be considered baseline values. For the peak number of eosinophils, hematoxylin and eosin stained esophageal biopsy specimen will be assessed and the high-powered fields with the highest density of eosinophils will be counted.
Proportion of patients with histological remission AND improvement in the dysphagia severity score from Baseline to end of treatment | From Baseline (Visit 2 + 3) to end of treatment (Visit 5 = 4-7 weeks after Visit 2)
  The processing and analysis of biopsy samples taken at Visit 2 and end of treatment (Visit 5) will be performed blinded at a central laboratory according to a laboratory manual. At both visits, 6 biopsy samples will be taken, 2 each from the proximal, mid, and distal segment of the esophagus. Additionally, patients will rate the dysphagia and odynophagia severity score daily on a 11-point NRS (numeric rating scale): 0 = 'no symptoms' to 10 = 'worst possible symptoms'. Patients will assess the severity score of the actual day in the patient diary daily after IMP intake starting on Day 0.
Absolute change in dysphagia and odynophagia severity scores from Baseline | From Baseline (Visit 3) to end of treatment (Visit 5 = 28 days after Visit 3)
  Patients will rate the dysphagia and odynophagia severity score daily on a 11-point NRS (numeric rating scale): 0 = 'no symptoms' to 10 = 'worst possible symptoms'. Patients will assess the severity score of the actual day in the patient diary daily after IMP intake starting on Day 0.
Relative change in dysphagia and odynophagia severity scores from Baseline | From Baseline (Visit 3) to end of treatment (Visit 5 = 28 days after Visit 3)
  Patients will rate the dysphagia and odynophagia severity score daily on a 11-point NRS (numeric rating scale): 0 = 'no symptoms' to 10 = 'worst possible symptoms'. Patients will assess the severity score of the actual day in the patient diary daily after IMP intake starting on Day 0.
Time to achieve symptom relief (defined as 50 percent improvement in the dysphagia or odynophagia symptoms on an NRS compared to Baseline) | From Baseline (Visit 3) to end of treatment (Visit 5 = 28 days after Visit 3)
  Patients will rate the dysphagia and odynophagia severity score daily on a 11-point NRS (numeric rating scale): 0 = 'no symptoms' to 10 = 'worst possible symptoms'. Patients will assess the severity score of the actual day in the patient diary daily after IMP intake starting on Day 0.
Change in the EREFS from Baseline to end of treatment | From Baseline (Visit 2) to end of treatment (Visit 5 = 4-7 weeks after Visit 2)
  The EREFS score (Eosinophilic esophagitis endoscopic reference score) is a classification and grading system for the endoscopic assessment of the esophageal features of eosinophilic esophagitis. The grading is used either to assess the severity of endoscopic findings from 0=´none´ to 2 or 3=´severe´ or to classify 0=´absent´ or 1=´present´.The total score will be calculated and compared between Baseline and end of treatment. A higher score correlates with more severe eosinophilic esophagitis symptoms.
Incidence of treatment-emergent Adverse Events | Visit 3 (Day 0) to day 42
  All Adverse Events occurring from the first investigational medicinal product administration onwards are defined as treatment-emergent Adverse Events.
Incidence of treatment-emergent Serious Adverse Events | Visit 3 (Day 0) to day 42
  All Serious Adverse Events occurring from the first investigational medicinal product administration onwards are defined as treatment-emergent Serious Adverse Events.
Incidence of AESI | Visit 2 (day -21 to -1) to Visit 6 (day 42)
  The following AEs are defined as AEs of special interest (AESI), if these events were not already present at Visit 2:
  * Oral candidiasis;
  * Oropharyngeal candidiasis.
Local tolerability | From Baseline (Visit 3) to end of treatment (Visit 5 = 28 days after Visit 3)
  The local tolerability of the IMP administration will be evaluated daily throughout the treatment period in the patient diary. Patients should indicate whether they had any discomfort in mouth, throat or esophagus while taking IMP on a VAS (Visual analog scale) ranging from 'no discomfort' to 'the worst imaginable discomfort'. The first assessment on Day 0 recorded in the patient diary after IMP intake will be considered Baseline.
Patient-reported treatment satisfaction at end of treatment based on questions about handling, taste, and time necessary for administration | At end of treatment (Visit 5 = day 28)
  Patients will be asked to answer a questionnaire about their satisfaction with the IMP treatment at Visit 5. Questions will cover the general satisfaction with the IMP, the swallowability of the IMP, and the frequency of administration. Answers involve gradings from 0 (the best outcome) to 3 or 4 (the worst outcome) plus an indication for the preference of single or multiple administrations of the investigated product.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Racamier, Study Director — EsoCap AG (Malzgasse 9, 4052 Basel, Switzerland)
Locations (17):
- Germany (4):
  - Facharztzentrum Eppendorf, Hamburg
  - Universitätsklinikum Leipzig AöR, Leipzig
  - Otto-von-Guericke-Universität Medizinische Fakultät Universitätsklinikum Magdeburg A. ö. R., Magdeburg
  - Klinikum rechts der Isar der TUM, München
- Netherlands (2):
  - Amsterdam University Medical Center, Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordrecht
- Poland (2):
  - Centrum Medyczne Med-GASTR Sp. z o.o., Lodz
  - Centrum Medyczne Sonomed Sp. z o.o., Szczecin
- Spain (8):
  - Hospital Universitario Vall d' Hebrón, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario Central De Asturias, Oviedo
  - Hospital de Navarra, Pamplona
  - Hospital General de Tomelloso, Tomelloso
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital de Viladecans, Viladecans
- Universitätsspital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lucendo AJ, Nantes-Castillejo O, Straumann A, Biedermann L, Bredenoord AJ, Guagnozzi D, Blas-Jhon L, Wiechowska-Kozlowska A, Weidlich S, von Arnim U, Santander-Vaquero C, Perello A, Perez-Martinez I, Barrio J, Vieth M, Gouya G, Dellon ES. Clinical Trial: Safety and Efficacy of a Novel Oesophageal Delivery System for Topical Corticosteroids Versus Placebo in the Treatment of Eosinophilic Oesophagitis. Aliment Pharmacol Ther. 2025 Feb;61(3):444-455. doi: 10.1111/apt.18443. Epub 2024 Dec 16. PMID 39676687